CLINICAL TRIAL: NCT00392795
Title: The BRAIN ICU Study: Bringing to Light the Risk Factors and Incidence of Neuropsychological Dysfunction in ICU Survivors
Brief Title: The BRAIN Intensive Care Unit (ICU) Study: Bringing to Light the Risk Factors
Acronym: BRAIN-ICU
Status: Active, not recruiting | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Wes Ely, Professor of Medicine, Vanderbilt University Medical Center
Other Study IDs: AG072472 01A1; R01AG027472 (NIH)
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Delirium; Cognition Disorders; Dementia
Keywords: Critical Care; Delirium; Long-term cognitive impairment; mechanical ventilation; Critical illness; dementia; sedatives and analgesics; aging
MeSH Terms: conditions — Delirium; Cognition Disorders; Dementia; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary purpose of this proposal will be to identify potentially modifiable risk factors of long-term cognitive impairment (i.e. development of delirium and exposure to sedative and analgesic medications) in ICU patients. The investigators will quantify the independent contribution of these risk factors to the incidence of long-term cognitive impairment, controlling for other established risk factors including age, pre-existing cognitive impairment, and apolipoprotein E (apoE) genotype. Quantifying the contributions of these modifiable risk factors will pave the way for the development of preventive and/or treatment strategies to reduce the incidence, severity and/or duration of long-term cognitive impairment and improve functional recovery for patients with critical illness.

DETAILED DESCRIPTION:
Among Intensive Care Unit (ICU) survivors, subsequent cognitive and functional decline are the greatest threats to meaningful recovery. Six small cohorts indicate that an alarming 30% to 80% of the increasingly millions of ICU survivors develop an acquired long-term cognitive impairment (LTCI) functionally equivalent to mild/moderate dementia that may last years. Additionally, major deficits in health-related quality of life (HRQL), functional status, and an "ICU accelerated" frailty are common, especially in the elderly. A leading and potentially modifiable risk factor for these devastating outcomes may be ICU delirium, which is a predictor of higher mortality, higher cost, and poor cognitive function at discharge. Additionally, heavy and prolonged exposure to potent psychoactive medications routinely administered in high doses to ventilated patients may have lasting yet preventable cognitive and functional effects. In this proposal, Aims 1 and 3 will determine whether delirium is an independent risk factor for the incidence, severity, and/or duration of LTCI (Aim 1) and impaired HRQL (Aim 3) in ICU survivors. Likewise, Aims 2 and 4 will determine whether degree of exposure to sedative and analgesic medications in ICU patients is an independent risk factor for the incidence, severity, and/or duration of LTCI (Aim 2) and impaired HRQL (Aim 4). The study will be a prospective cohort study enrolling 800 mechanically ventilated medical and surgical patients from 3 diverse medical centers over a 39 month period with comprehensive follow-up testing at 3 and 12 months after hospital discharge. This study will quantify whether delirium and sedative/analgesic exposure are indeed risk factors for LTCI and HRQL, controlling for other covariates such as age, medical versus surgical ICU admission, pre-existing cognitive impairment, sepsis, and apoE genotype. This will pave the way for the development of preventive and/or treatment strategies to reduce long-term cognitive impairment and improve the functional recovery of older and younger ICU patients for decades to come. Major threats to recovery for ICU survivors are acquired cognitive and functional decline that can last years, especially in older patients. To pave the way for future preventive and interventional strategies, the cohort will determine to what degree delirium and potent sedatives and analgesics are risk factors for long-term cognitive impairment and functional decline following critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if they are adult, patients in a medical and/or surgical ICU receiving treatment for any of the following: respiratory failure or cardiogenic or septic shock.

Exclusion Criteria:

Patients who meet the inclusion criteria will be excluded if they meet any of the following criteria:

* Cumulative ICU time >5 days in the past 30 days, not including the current ICU stay, as this might create a state of flux regarding patients' cognitive baseline
* Severe cognitive or neurodegenerative diseases that prevent a patient from living independently at baseline, including mental illness requiring institutionalization, acquired or congenital mental retardation, known brain lesions, traumatic brain injury, cerebrovascular accidents with resultant moderate to severe cognitive deficits or ADL dependency, Parkinson's disease, Huntington's disease, severe Alzheimer's disease or dementia of any etiology
* ICU admission post cardiopulmonary resuscitation with suspected anoxic injury
* An active substance abuse or psychotic disorder, or a recent (within the past 6 months) serious suicidal gesture necessitating hospitalization. This exclusion will enrich follow-up rates by avoiding patients with whom it is particularly challenging to maintain long-term contact
* Blind, deaf, or unable to speak English, as these conditions would preclude our ability to perform the follow-up evaluation interviews.
* Overly moribund and not expected to survive for an additional 24 hours and / or withdrawing life support to focus on comfort measures only.
* Prisoners.
* Patients who live further than 200 miles from Nashville and who do not regularly visit the Nashville area.
* Patients who are homeless and have no secondary contact person available. This exclusion will enrich follow-up rates by avoiding patients with whom it is particularly challenging to maintain long-term contact
* The onset of the current episode of respiratory failure, cardiogenic shock, or septic shock was > 72 hours ago.
* Patients who have had cardiac bypass surgery within the past 3 months (including the current hospitalization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Medical and Surgical ICUs
Sampling Method: Probability Sample
Enrollment: 826 (Actual)
Dates: Start 2007-01; Primary Completion 2010-12 (Actual); Study Completion 2026-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: E Wesley Ely, MD, MPH, Principal Investigator — Vanderbilt University/VA TN Valley GRECC
Locations (2):
- United States (2):
  - Saint Thomas Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee

REFERENCES:
- [Background] Ely EW, Shintani A, Truman B, Speroff T, Gordon SM, Harrell FE Jr, Inouye SK, Bernard GR, Dittus RS. Delirium as a predictor of mortality in mechanically ventilated patients in the intensive care unit. JAMA. 2004 Apr 14;291(14):1753-62. doi: 10.1001/jama.291.14.1753. PMID 15082703
- [Background] Ely EW, Truman B, Shintani A, Thomason JW, Wheeler AP, Gordon S, Francis J, Speroff T, Gautam S, Margolin R, Sessler CN, Dittus RS, Bernard GR. Monitoring sedation status over time in ICU patients: reliability and validity of the Richmond Agitation-Sedation Scale (RASS). JAMA. 2003 Jun 11;289(22):2983-91. doi: 10.1001/jama.289.22.2983. PMID 12799407
- [Background] Ely EW, Inouye SK, Bernard GR, Gordon S, Francis J, May L, Truman B, Speroff T, Gautam S, Margolin R, Hart RP, Dittus R. Delirium in mechanically ventilated patients: validity and reliability of the confusion assessment method for the intensive care unit (CAM-ICU). JAMA. 2001 Dec 5;286(21):2703-10. doi: 10.1001/jama.286.21.2703. PMID 11730446
- [Background] Jackson JC, Gordon SM, Ely EW, Burger C, Hopkins RO. Research issues in the evaluation of cognitive impairment in intensive care unit survivors. Intensive Care Med. 2004 Nov;30(11):2009-16. doi: 10.1007/s00134-004-2422-2. Epub 2004 Sep 15. PMID 15372146
- [Background] Jackson JC, Gordon SM, Hart RP, Hopkins RO, Ely EW. The association between delirium and cognitive decline: a review of the empirical literature. Neuropsychol Rev. 2004 Jun;14(2):87-98. doi: 10.1023/b:nerv.0000028080.39602.17. PMID 15264710
- [Background] Ely EW, Wheeler AP, Thompson BT, Ancukiewicz M, Steinberg KP, Bernard GR. Recovery rate and prognosis in older persons who develop acute lung injury and the acute respiratory distress syndrome. Ann Intern Med. 2002 Jan 1;136(1):25-36. PMID 11777361
- [Background] Ely EW, Evans GW, Haponik EF. Mechanical ventilation in a cohort of elderly patients admitted to an intensive care unit. Ann Intern Med. 1999 Jul 20;131(2):96-104. doi: 10.7326/0003-4819-131-2-199907200-00004. PMID 10419447
- [Background] Hopkins RO, Weaver LK, Pope D, Orme JF, Bigler ED, Larson-LOHR V. Neuropsychological sequelae and impaired health status in survivors of severe acute respiratory distress syndrome. Am J Respir Crit Care Med. 1999 Jul;160(1):50-6. doi: 10.1164/ajrccm.160.1.9708059. PMID 10390379
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Derived] Rengel KF, Wilson JE, Silver HJ, Hollingsworth E, Orun OM, Jackson JC, Mart MF, Hughes CG, Ely EW, Brummel NE. Associations Among Skeletal Muscle Health, Disability, and Self-Reported Physical Function in Survivors of Critical Illness: A Secondary Analysis of the Bringing to Light the Risk Factors and Incidence of Neuropsychological Dysfunction in ICU Survivors Study. CHEST Crit Care. 2025 Jun;3(2):100115. doi: 10.1016/j.chstcc.2024.100115. Epub 2024 Nov 29. PMID 40837197
- [Derived] Hughes CG, Hayhurst CJ, Pandharipande PP, Shotwell MS, Feng X, Wilson JE, Brummel NE, Girard TD, Jackson JC, Ely EW, Patel MB. Association of Delirium during Critical Illness With Mortality: Multicenter Prospective Cohort Study. Anesth Analg. 2021 Nov 1;133(5):1152-1161. doi: 10.1213/ANE.0000000000005544. PMID 33929361
- [Derived] Duggan MC, Morrell ME, Chandrasekhar R, Marra A, Frimpong K, Nair DR, Girard TD, Pandharipande PP, Ely EW, Jackson JC. A Brief Informant Screening Instrument for Dementia in the ICU: The Diagnostic Accuracy of the AD8 in Critically Ill Adults Suspected of Having Pre-Existing Dementia. Dement Geriatr Cogn Disord. 2019;48(5-6):241-249. doi: 10.1159/000490379. Epub 2020 Apr 7. PMID 32259825
- [Derived] Hayhurst CJ, Patel MB, McNeil JB, Girard TD, Brummel NE, Thompson JL, Chandrasekhar R, Ware LB, Pandharipande PP, Ely EW, Hughes CG. Association of neuronal repair biomarkers with delirium among survivors of critical illness. J Crit Care. 2020 Apr;56:94-99. doi: 10.1016/j.jcrc.2019.12.010. Epub 2019 Dec 16. PMID 31896448
- [Derived] Wilson JE, Duggan MC, Chandrasekhar R, Brummel NE, Dittus RS, Ely EW, Patel MB, Jackson JC. Deficits in Self-Reported Initiation Are AssociatedWith Subsequent Disability in ICU Survivors. Psychosomatics. 2019 Jul-Aug;60(4):376-384. doi: 10.1016/j.psym.2018.09.004. Epub 2018 Sep 29. PMID 30352696
- [Derived] Hayhurst CJ, Jackson JC, Archer KR, Thompson JL, Chandrasekhar R, Hughes CG. Pain and Its Long-term Interference of Daily Life After Critical Illness. Anesth Analg. 2018 Sep;127(3):690-697. doi: 10.1213/ANE.0000000000003358. PMID 29649027
- [Derived] Brummel NE, Bell SP, Girard TD, Pandharipande PP, Jackson JC, Morandi A, Thompson JL, Chandrasekhar R, Bernard GR, Dittus RS, Gill TM, Ely EW. Frailty and Subsequent Disability and Mortality among Patients with Critical Illness. Am J Respir Crit Care Med. 2017 Jul 1;196(1):64-72. doi: 10.1164/rccm.201605-0939OC. PMID 27922747
- [Derived] Jackson JC, Pandharipande PP, Girard TD, Brummel NE, Thompson JL, Hughes CG, Pun BT, Vasilevskis EE, Morandi A, Shintani AK, Hopkins RO, Bernard GR, Dittus RS, Ely EW; Bringing to light the Risk Factors And Incidence of Neuropsychological dysfunction in ICU survivors (BRAIN-ICU) study investigators. Depression, post-traumatic stress disorder, and functional disability in survivors of critical illness in the BRAIN-ICU study: a longitudinal cohort study. Lancet Respir Med. 2014 May;2(5):369-79. doi: 10.1016/S2213-2600(14)70051-7. Epub 2014 Apr 7. PMID 24815803
- [Derived] Pandharipande PP, Girard TD, Jackson JC, Morandi A, Thompson JL, Pun BT, Brummel NE, Hughes CG, Vasilevskis EE, Shintani AK, Moons KG, Geevarghese SK, Canonico A, Hopkins RO, Bernard GR, Dittus RS, Ely EW; BRAIN-ICU Study Investigators. Long-term cognitive impairment after critical illness. N Engl J Med. 2013 Oct 3;369(14):1306-16. doi: 10.1056/NEJMoa1301372. PMID 24088092
- See also: ICU Delirium and Cognitive Impairment Study Group Website — http://www.icudelirium.org